CLINICAL TRIAL: NCT06224673
Title: Phase II Open-label Study of ARX788 (Anti-HER2 Antibody Drug Conjugate (ADC)) for Patients With HER2-low Locally Advanced Unresectable or Metastatic Breast Cancer
Brief Title: ARX788 for Treating Patients With HER2-low Locally Advanced Unresectable or Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Laura Huppert, MD, BA (Other)
Collaborators: Ambrx, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Laura Huppert, MD, BA, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 237527; NCI-2024-00073 (Registry Identifier: University of California, San Francisco)
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: HER2 Low Breast Carcinoma; Triple Negative Breast Cancer; Hormone-receptor-positive Breast Cancer; Hormone Receptor Positive Breast Carcinoma
Keywords: Antibody-drug Conjugate
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ARX788; Specimen Handling; Amiloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: HR+/HER2-low (Experimental): Participants with locally advanced, unresectable MBC that is hormone receptor (HR) positive (HR+) /human epidermal growth factor receptor 2 (HER2)-low will receive ARX788 intravenously over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants also undergo CT, PET/CT, and collection of blood samples throughout the study.
  Interventions: Drug: ARX788; Procedure: Computed Tomography (CT); Procedure: Biospecimen Collection
- Cohort 2: HR-/HER2-low (Experimental): Participants with confirmed HR negative (HR-)/human epidermal growth factor receptor 2 (HER2)-low will receive ARX788 intravenously over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. Participants also undergo CT, PET/CT, and collection of blood samples throughout the study.
  Interventions: Drug: ARX788; Procedure: Computed Tomography (CT); Procedure: Biospecimen Collection
- Ocular Toxicity Prevention Sub-study (Experimental): The first 5 participants from Cohorts 1 and 2 will be given outpatient eye drops to use from home in conjunction with ARX788. Participants will be drop applied to each eye 4 times a day starting on the day of first infusion and continuing daily throughout treatment and for 30 days after the last infusion.
  Interventions: Drug: ARX788; Procedure: Computed Tomography (CT); Procedure: Biospecimen Collection; Drug: Amiloride

INTERVENTIONS:
Drug: ARX788 — Given IV
  Other Names: Anvatabart Opadotin; Antibody-drug Conjugate ARX788; Anti-Her2 Mab PAF- MMAF Toxin Oxime Conjugate ARX-788; Anti-Her2 ADC
Procedure: Computed Tomography (CT) — Undergo CT or Positron Emission Tomography(PET)/CT
  Other Names: CT Scan; PET/CT
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Specimen Collection; Biological Sample Collection
Drug: Amiloride — Ophthalmologic drops given topically to participants for an eye toxicity substudy
  Other Names: Amiloride Topical Eye Drops
  Arms: Ocular Toxicity Prevention Sub-study

SUMMARY:
This phase II trial tests how well ARX788 works in treating patients diagnosed with HER2-low, locally advanced unresectable or metastatic breast cancer. ARX788 is an antibody-drug conjugate (ADC) that is given by infusion (diluted and injected slowly into veins). Antibodies are proteins which are naturally produced by the body's immune system to help fight infections. ARX788 consists of antibodies that have been attached to a toxin that has the potential to kill cancer cells. ARX788 sticks to a protein called human epidermal growth factor receptor (HER2), which is found on some breast cancer cells. Giving ARX788 may be safe and effective in treating patients with HER2-low locally advanced unresectable metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the objective response rate (ORR) of participants with HER2-low locally advanced unresectable/metastatic breast cancer on ARX788 monotherapy.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of ARX788 monotherapy in participants with HER2-low locally advanced unresectable or metastatic breast cancer (MBC) as measured by duration of response (DOR), best overall response (BOR), disease control rate (DCR), progression-free survival (PFS), and overall survival (OS).

II. To evaluate the safety of ARX788 monotherapy in participants with HER2-low locally advanced unresectable or MBC.

III. To evaluate the safety, tolerability, adherence, and feasibility of the eye toxicity prevention regimen in the ocular toxicity prevention sub study.

IV. To evaluate the efficacy of the eye toxicity prevention regimen in the ocular toxicity prevention sub study.

EXPLORATORY OBJECTIVES:

I. Biomarker analyses to evaluate association of efficacy measures with potential biomarkers (e.g., via assessment of circulating tumor deoxyribonucleic acid (ctDNA), single cell ribonucleic acid (RNA) sequencing, etc.).

II. Patient-reported outcomes (PROs) of patients on ARX788 monotherapy.

III. To determine the pharmacokinetics (PK) of ARX788 in tears.

OUTLINE:

Participants are assigned to cohorts based on breast cancer subtype and receive ARX788 intravenously (IV) over 90 minutes on day 1 of each cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity. The first 5 participants successfully enrolled will receive topical amiloride 0.1% to evaluate early safety, tolerability, adherence, and feasibility data. Participants may continue study treatment until progressive disease, intolerable side effects, discontinuation due to Investigator's clinical judgment, discontinuation due to patient's choice, or the Sponsor-investigator's decision to stop the study. After completion of study treatment, participants are followed up at 30 days and then every 12 weeks for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants age 18 years or greater with ability to provide written informed consent for the study.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2.
* Estimated life expectancy of at least at 6 months per investigator assessment.
* Ability to understand and the willingness to sign a written informed consent document.
* Pathologically documented HER2-low locally advanced unresectable or metastatic breast cancer (MBC). NOTE: human epidermal growth factor receptor 2 (HER2)-low status determined by HER2 immunohistochemistry (IHC) 1+ or 2+ and no evidence of HER2 gene amplification by in situ hybridization (ISH)/fluorescence in situ hybridization (FISH), which can be documented from any tumor sample during the patient's cancer treatment history (early-stage or metastatic).

  * Cohort 1: Participants with hormone receptor positive (HR+)/HER2-low locally advanced unresectable or MBC. HR+ status defined as estrogen receptor >= 10% and/or progesterone receptor ≥ 10% and HER2 low.
  * Cohort 2: Participants with hormone receptor negative (HR-)/HER2-low locally advanced unresectable or MBC. Considered HR- if estrogen receptor (ER) and progesterone receptor (PR) < 10% and HER2-low.
* Presence of at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. NOTE: Participant's with at least one measurable lytic bone lesion are eligible.
* Availability of tumor block or formalin-fixed paraffin-embedded (FFPE) tissue as 10 precut unstained slides will be collected for the HER2 status evaluation and biomarker analysis based on the most recent tumor tissue sample. NOTE: New pretreatment biopsy tissue is preferred as HER2 status may change, but a fresh biopsy is not required. The study team and investigator will make every attempt to get archival tissue. Participants who do not have archival or new tumor tissue available may be eligible after discussion with the study principal investigator (PI).
* Participants with stable and treated brain metastases are eligible if the participants meet the following criteria:

  * Prior stereotactic radiosurgery (SRS) should be completed >=7 days before study treatment initiation.
  * Prior whole-brain radiation therapy should be completed >=14 days before study treatment initiation.
  * Any ongoing use of systemic corticosteroids does not exceed 2 mg of dexamethasone (or equivalent) daily.
* Participants must have received at least one prior line of chemotherapy or ADC therapy for locally advanced unresectable or metastatic disease. Prior checkpoint inhibitor therapy is allowed.
* Hemoglobin ≥ 8.0 g/dL
* Absolute neutrophil count ≥ 1.0 x 10^9/L
* Platelets ≥ 100,000 x 10^9/L
* Total bilirubin ≤ 1.5 x institutional upper limit of normal, unless elevated due to Gilbert's syndrome and direct bilirubin is within normal limits
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase (SGOT)) < 3 x institutional upper limit of normal. In participants with liver metastases, <= 5 x institutional upper limit of normal is allowed.
* Alanine aminotransferase (ALT) (serum glutamic-pyruvic transaminase (SGPT)) < 3 x institutional upper limit of normal. In participants with liver metastases, <=5 x institutional upper limit of normal is allowed.
* Creatinine ≤ 1.5 x within institutional upper limit of normal OR creatinine clearance glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m, calculated using the Cockcroft-Gault equation
* Adequate cardiac function as assessed by left ventricular ejection fraction ≥ 50% or institutional lower limit of normal.
* Human immunodeficiency virus (HIV)-infected individuals on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For participants with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy.
* Individuals with a history of hepatitis C virus (HCV) infection must have been treated without detectable HCV RNA.
* Participants must have recovered from all acute toxicities from prior therapies to ≤ grade 1 or baseline (except for alopecia and neuropathy) per the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) v 5.0.
* Male and female subjects of reproductive/childbearing potential must agree to use a highly effective form of contraception or total sexual abstinence during and upon completion of the study; and for at least 3 months after the last dose of study drug for women of childbearing potential (WOCBP) and at least 5 months after the last dose of study drug for men whose partners are WOCBP.
* Male subjects must agree to not freeze or donate sperm starting at Screening and throughout the study period, and at least 5 months after the final study drug administration.
* Female subjects must agree to not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 3 months after the final study drug administration.

Exclusion Criteria:

* Has a prior history of treatment with ARX-788 or auristatin analogues.
* Has a history of allergic reaction to any component of ARX788.
* Has exposure to any other investigational or commercial anti-cancer agents or therapies administered with the intention to treat malignancy within 14 days before the first dose of study treatment. NOTE: Anti-hormonal therapy may be administered up to 7 days prior to the first dose of study treatment.
* Radiotherapy outside of the brain administered <7 days prior to first dose of ARX788
* Prior or current history of interstitial lung disease (ILD), pneumonitis, or other clinically significant lung disease with the exception of disease that is directly attributable to the presence of lung metastases from their underlying cancer.
* Participants with significant pulmonary conditions, defined as any of the following:

  * Any prior history of drug-induced immune-mediated pneumonitis.
  * Prior history of radiation therapy to the chest of > 18 gray (Gy) with residual sequelae considered clinically significant by investigator assessment.
  * Radiographic evidence of radiation fibrosis involving > 15% of the lung parenchyma associated with clinical symptoms.
  * Any requirement for supplemental oxygen.
* Clinically-significant ocular findings including history of keratitis, keratopathy, and/or active eye disease (excluding glaucoma).
* History of congestive heart failure, unstable angina pectoris, unstable cardiac arrhythmia, or myocardial infarction within 6 months prior to enrollment. QTcF prolongation of >470 msec (females) or >450 msec (males) based screening ECG.
* Has a diagnosis of leptomeningeal carcinomatosis. NOTE: Stable brain metastases are allowed.
* Has an active systemic or psychiatric illness that would impact the patient's ability to receive study therapy.
* Has an uncontrollable intercurrent illness, infection (including participants with active, symptomatic Coronavirus disease of 2019 (COVID-19) infections), or other conditions that could limit study compliance or interfere with study assessments.
* Has a history of an additional malignancy that is progressing or has required active treatment within the past 3 years. NOTE: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ (excluding carcinoma in situ of the bladder or high-grade cervical dysplasia in the last three years), and thyroid cancer not requiring cytotoxic agents that have undergone potentially curative therapy are not excluded.
* Pregnancy or breastfeeding.
* Has an active, uncontrolled hepatitis B, hepatitis C, and/or human immunodeficiency virus (HIV) infection. Participants with adequately controlled hepatitis B, hepatitis C, and/or HIV are allowed. NOTE: HIV and hepatitis B and C testing are not required for screening. Testing will only be done if clinically indicated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-12-18 (Actual); Primary Completion 2029-03-31 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 1 year
  Objective response rate (ORR) is defined as the proportion of participants who experience complete response (CR) or partial response (PR) using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The ORR and corresponding two-sided exact 90% confidence intervals will be reported.

SECONDARY OUTCOMES:
Duration of response (DOR) | Up to 1 year
  Duration of response (DOR) is defined as the time between the date of first response and the date of disease progression or death, whichever occurs first, will be computed for participants with a BOR of CR or PR. Medians and corresponding two-sided 95% confidence intervals will be reported.
Overall Best Response (BOR) | Up to 1 year
  Best overall response (BOR) is defined as the best response recorded from the start of the treatment until disease progression (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
Disease Control Rate (DCR) | Up to 1 year
  The Disease control rate (DCR) is defined as the sum of PR, CR and stable disease (SD) divided by the number of response evaluable participants All-Subjects-as-Treated(AsaT).
Median Progression Free Survival (PFS) | Up to 2 years
  Progression-free survival (PFS) is defined as the time between date of first dose of study therapy and date of progression or death, whichever occurs first, will be computed for response evaluable participants (AsaT). Medians and corresponding two-sided 95% confidence intervals will be reported.
Median Overall Survival (OS) | Up to 2 years
  Overall survival (OS) is defined as the amount of time that elapses between the initiation of therapy (Cycle 1, Day 1 (C1D1) and the time of death from any cause. Medians and corresponding two-sided 95% confidence intervals will be reported.
Proportion of participants with treatment-emergent adverse events (AEs) | Up to 1 year
  Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.
Percentage of participants adhering to the eye drop | Up to 1 year
  Tolerability and adherence to eye toxicity prevention regimen will be reported as the percentage of participants who adhered to the regimen during the course of the study.
Mean score on an eye pain scale | Up to 1 year
  After each drop, participants will assess the amount of pain on a scale from 1 (lowest amount) to 10 (greatest amount). The mean and standard deviation of the pain scores by cohort will be reported
Proportion of participants reporting ocular adverse events | Up to 1 year
  The proportion of participants with a recorded grade >=2 ocular AEs based on visual acuity, eye symptoms, cornea evaluation and intraocular pressure (mmHg) readings will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Huppert, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No